CLINICAL TRIAL: NCT06567990
Title: Type 2 DIAbeTes With NAFLD: innOvative Biomarkers of Disease progressioN and clInical outComes
Acronym: DIATONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 69HCL24_0022
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Dysfunction-Associated Liver Disease
Keywords: MASLD; Type 2 diabetes; Obesity; Advanced fibrosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, multi-site, not randomized, national study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with T2D and MASLD without advanced fibrosis (AF) (COHORT A) (Other): Patients with T2D and MASLD without advanced fibrosis (AF) at baseline in the NAFLD-Care study.
  Interventions: Diagnostic Test: Non-invasive test for the screening of MASLD-related advanced fibrosis in patients with T2D.
- Patients with T2D and MASLD, without diagnosis of cirrhosis (COHORT B) (Other): Patients with T2D and MASLD with presence of advanced fibrosis (AF) and without cirrhosis at baseline in the NAFLD-Care study
  Interventions: Diagnostic Test: Non-invasive test for the screening of MASLD-related advanced fibrosis in patients with T2D.

INTERVENTIONS:
Diagnostic Test: Non-invasive test for the screening of MASLD-related advanced fibrosis in patients with T2D. — * Non-invasive blood biological tests = NAFLD Fibrosis Score, FIB-4 score, FNI score, Agile3+ score, FASTscore, ELF, Fibrotest, Fibrometer if performed in clinical care
  * Non-invasive imaging = Transient elastography (FibroScan), Questionnaire assessing alcohol consumption

SUMMARY:
Type 2 diabetes (T2DM) patients are at high-risk for advanced fibrosis (AF) due to non-alcoholic fatty liver disease (NAFLD), recently renamed Metabolic dysfunction-Associated Liver Disease (MASLD). Thus, patients with T2DM are recognized as a priority target for the screening of MASLD-related advanced fibrosis and a systematic screening for AF is currently recommended in T2DM patients using FIB-4 and liver stiffness measurement (LSM).The main objective of the project is to investigate the ability of baseline non-invasive biomarkers to discriminate patients with a progression of MASLD from patients without progression of MASLD among patients with T2DM and to investigate the association between clinical outcomes related to the natural evolution of MASLD and T2DM and baseline biomarkers.

DETAILED DESCRIPTION:
Type 2 diabetes (T2DM) patients are at high-risk for advanced fibrosis (AF) due to non-alcoholic fatty liver disease (NAFLD), recently renamed Metabolic dysfunction-Associated Liver Disease (MASLD). Thus, patients with T2DM are recognized as a priority target for the screening of MASLD-related advanced fibrosis and a systematic screening for AF is currently recommended in T2DM patients using FIB-4 and liver stiffness measurement (LSM). Hence, these Non-Invasive Tests (NITs) are expected to be integrated in the management of T2DM in a near future. Indeed diabetologists are becoming more aware of the need for liver assessment in patients with T2DM recently reinforced by recent clear recommendations supporting the use of non-invasive test (NITs) such as LSM for the detection of liver fibrosis. Several studies indicate that MASLD increases the risk of T2DM complications. However, there are very limited data and no prospective longitudinal data assessing the progression of MASLD and relevant clinical outcomes in T2DM patients included in liver screening using these NITs. This provides a unique opportunity to better stratify T2DM and to understand the heterogeneity among patients with T2DM by defining patient's profiles linked the progression of MASLD and relevant clinical outcomes.

Therefore, the main objective of the project is to investigate the ability of baseline non-invasive biomarkers to discriminate patients with a progression of MASLD from patients without progression of MASLD among patients with T2DM and to investigate the association between clinical outcomes related to the natural evolution of MASLD and T2DM and baseline biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2D and meeting the other inclusion criteria of the NAFLD-Care study:
* Patient aged between 40 and 80 years old,
* Patient with hepatic steatosis determined by conventional abdominal ultrasound as defined by the EASL/EASO/EASD European guidelines.
* Patient who agrees to be included in the study and who signs the informed consent form,
* Patient affiliated to a healthcare insurance plan.

Exclusion Criteria:

- Participants with a diagnosis of cirrhosis defined by a liver biopsy with histological stage of fibrosis F4 or a proven diagnosis of cirrhosis by magnetic resonance imaging.

The main non-inclusion criteria for the NAFLD-CARE study are:

* Evidence of other causes of chronic liver disease :

  1. Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
  2. Previous or current infection with Hepatitis C as defined by presence of hepatitis C virus Ab in serum (anti-HCV Ab).
  3. Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
  4. Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
  5. Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
  6. Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
  7. Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
  8. Drug-induced liver disease as defined on the basis of typical exposure and history.
  9. Bile duct obstruction as shown by imaging studies.
* History of ingestion of medications known to produce steatosis in the previous 6 months.
* Evidence of cirrhosis or previously known cirrhosis based on the results from previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy or varices
* Presence of regular and/or excessive use of alcohol (defined as >30g/day for males and >15g/day for females) for a period longer than 2 years at any times in the last 10 years
* The subject is a pregnant or nursing female
* Life expectancy less than 5 years
* History of known HIV infection
* History of type 1 diabetes
* BMI ≥ 45 kg/m2
* Mentally unbalanced patients, under supervision or guardianship,
* Patient deprived of liberty,
* Patient who does not understand French/ is unable to give consent,
* Patient already included in a trial who may interfere with the study or in a period of exclusion following participation in a previous study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Progression of MASLD for T2D and MASLD patients without AF at baseline (cohort A) or progression to confirmed diagnosis of cirrhosis for T2D and MASLD patients with presence of AF at baseline and without cirrhosis (cohort B). | One time visit planned according to standard care at 4 years+/- 6 months after inclusion in the NAFLD-CARE study
  COHORT A = Composite outcome defined by either histological stage of fibrosis ≥ F3 if a liver biopsy is performed in clinical care or concordant patented Fibrotest≥ F3 and LSM≥ 8 kPa according to EASL guidelines or overt imaging evidence of cirrhosis via ultrasound, computed tomography (CT), or MRI COHORT B = Histological stage of fibrosis 4 or imaging evidence of cirrhosis via ultrasound, computed tomography (CT), or MRI

SECONDARY OUTCOMES:
Assessment of clinical events associated with the natural history of MASLD and T2D for both cohorts | One time visit planned according to standard care at 4 years+/- 6 months after inclusion in the NAFLD-CARE study
  Occurrence of T2D COMPLICATIONS (retinopathy, neuropathy, nephropathy, diabetes foot ulcer ), CARDIOVASCULAR EVENTS (coronary artery disease, myocardial infarction, coronary revascularization, stroke, arteriopathy of the lower limbs), LIVER RELATED EVENTS (ascites, esophageal variceal bleeding or needed prophylactic treatment, liver transplantation, hepatocellular carcinoma), KIDNEY RELATED EVENTS (occurence or progression of diabetic nephropathy), DEATHS (all causes).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service Endocrinologie, Diabétologie, Maladies Métaboliques et Nutrition, Dijon
  - Endocrinologie, Diabète et Nutrition in Louis PRADEL Hospital, Lyon
  - Clinique d'Endocrinologie, Maladies Métaboliques et Nutrition CIC Endocrino-Nut, Nantes
  - Service d'Endocrinologie, Diabète et nutrition, Pierre-Bénite